CLINICAL TRIAL: NCT01189526
Title: A Randomized Trial Comparing Intravitreal Ranibizumab and Macular Laser Photocoagulation for the Treatment of Macular Edema Following Branch Retinal Vein Occlusion
Brief Title: Comparison of Intravitreal Ranibizumab and Macular Laser Photocoagulation for ME Following Branch Retinal Vein Occlusion (BRVO)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul Retina Investigator Group (Network)
Collaborators: Samsung Medical Center (Other); Kyungpook National University Hospital (Other)
Responsible Party: Se Woong Kan, M.D. and Jae Pil Shin, M.D., Samsung Medical Center and Kyungpook National University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RVOIVRI; BRVOIVRI
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Last update posted 2010-08-26 (Estimated); Status verified 2010-08

CONDITIONS: Branch Retinal Vein Occlusion
Keywords: Branch retinal vein occlusion; macular edema; intravitreal injection; ranibizumab
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVRI (Experimental): IVRI : intravitreal ranibizumab (0.5mg) injection
  Interventions: Drug: Ranibizumab
- Laser (Active Comparator): Laser : macular laser photocoagulation
  Interventions: Procedure: macular laser photocoagulation

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab 0.5mg Ranibizumab will be administered to patients as multiple intravitreal injections.
  Arms: IVRI
Procedure: macular laser photocoagulation — Treatment may include both focal and grid therapy using the laser and contact lens of the investigator's choice.
  Arms: Laser

SUMMARY:
This study is designed to evaluate the efficacy of intravitreal Ranibizumab in comparison with macular laser photocoagulation as treatments for macular edema secondary to branch retinal vein occlusion.

Characteristics of this study is as below

1. Multicenter, randomized clinical trial. (intravitreal Ranibizumab 0.5mg injection vs. macular laser photocoagulation)
2. After 48 weeks follow up, functional change(visual acuity)and anatomical change (central retinal thickness) would be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Symptom duration < 6 Months, > 4 weeks
* Visual acuity - less than 20/40 (73 letters) more than 20/400 (19 letters) in ETDRS chart
* OCT - center involved retinal thickening : > 250 micrometers
* clear media
* well controlled hypertension (<140/90mmHg) and diabetes (6.5<HbA1c<9.5)
* willing to return for all scheduled visits

Exclusion Criteria:

* uveitis,NVG, exudative AMD, diabetic retinopathy, Irvine-Gass syndrome, OIS
* any malignancy
* previous treatment history - laser photocoagulation, intravitreal injection with any drug, vitrectomy
* vitreomacular traction or epiretinal membrane
* intraocular surgery in the study eye within 6 months
* uncontrolled glaucoma ( > 30mmHg with anti-glaucoma medications)
* optic neuropathy, amblyopia
* A condition that in the opinion of the investigator would preclude a patient's participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (ETDRS letters) | 48 weeks

SECONDARY OUTCOMES:
Retinal Thickening | 48 weeks
  Optical Coherence Tomography measured central retinal thickness

CONTACTS AND LOCATIONS:
Overall Officials: Se Woong Kang, M.D., Principal Investigator — Department of Ophthalmology, Samsung Medical Center, Sungkyunkwan University School of Medicine; Jae Pil Shin, M.D., Principal Investigator — Department of Ophthalmology, Kyungpook National University
Locations (1):
- Samsung Medical Center, Seoul, South Korea